CLINICAL TRIAL: NCT02511834
Title: VEST III PMS Clinical Protocol
Acronym: VEST III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD0113
Record Dates: First submitted 2015-07-25; First posted 2015-07-30 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VEST supported (Experimental): Vein graft supported by VEST
  Interventions: Device: VEST External Support; Procedure: Coronary Artery Bypass Surgery
- Control (Active Comparator): Vein grafts unsupported by VEST
  Interventions: Procedure: Coronary Artery Bypass Surgery

INTERVENTIONS:
Device: VEST External Support
  Arms: VEST supported
Procedure: Coronary Artery Bypass Surgery
  Other Names: CABG

SUMMARY:
Post marketing surveillance (PMS) study. 200 patients will be enrolled in a prospective, multi center, randomized, two-arm, open label, and controlled, enrolling patients with multi vessel atherosclerotic coronary artery disease, scheduled to undergo Coronary artery bypass grafting (CABG) with arterial grafting of IMA to LAD, one saphenous vein graft (SVG) to the right territory and one or more SVGs to the left territory. Of all vein grafts, one will be selected randomly to receive treatment with VEST and another designated Control.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for on-pump CABG on clinical grounds
2. Two or more bypass vein grafts bypasses indicated as follows: one (1) for right coronary artery, 1 or more for left coronary arteries and IMA indicated for the LAD on clinical grounds
3. Appropriately sized and accessible target coronary arteries, with a minimum diameter of 1.5 mm and adequate vascular bed
4. Ability to give their informed written consent
5. Ability and willingness to comply with study follow up requirements
6. Patient is ≥ 18 and ≤ 80 years of age, and has Life expectancy ≥5 years

Exclusion Criteria:

1. Concomitant non-CABG cardiac procedure
2. Prior cardiac surgery
3. Emergency CABG surgery (cardiogenic shock, inotropic pressure support, IABP)
4. Contraindication for on-pump CABG with cardioplegic arrest (e.g. severely calcified aorta)
5. Calcification at the intended anastomotic sites, as assessed upon opening of the chest, before randomization
6. Severe vein varicosity
7. Prior debilitating stroke less than 1 year before surgery
8. Severe renal dysfunction (Cr>2.0 mg/dL or >177 μmol/L)
9. Women of child bearing age
10. Concomitant life-threatening disease likely to limit life expectancy to less than 5 years
11. Indication for Warfarin up to time of surgery
12. Inability to tolerate or comply with required normal post-operative drug regimen (antiplatelet, statin and beta-blockers) that cannot adequately be controlled.
13. inability to take aspirin
14. Contraindication to intravascular contrast material that cannot be adequately controlled with pre-medication
15. Inability to comply with required follow-ups including angiographic and/or CT imaging methods.
16. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Proportion of Vein grafts with Fitzgibbon I patency score out of all grafts including occluded ones. | 2 years
  Perfect patency, no lumen irregularities. Rates out of all grafts including occluded ones.

SECONDARY OUTCOMES:
Intimal hyperplasia area | 2 years
  Sub group (IVUS) - Intimal hyperplasia (plaque+media) area [mm2] as assessed by IVUS
MACCE | 2 years
  Composite of: All-cause mortality; Stroke; Myocardial infarction; Coronary revascularization
Vein graft failure | 2 years
  Defined as ≥50% stenosis by QCA
Early vein graft failure | 6 months
  Early vein graft failure, defined as >50% occlusion by CT Angio

CONTACTS AND LOCATIONS:
Locations (15):
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Medical University of Vienna, Vienna
- Germany (6):
  - German Heart Center, Berlin
  - Immanuel Hospital Bernau. Brandenburg Heart Center, Bernau
  - University Hospital of Cologne, Cologne
  - West-German Heart Center Essen University, Essen
  - University Medical Center Schleswig-Holstein, Lübeck
  - Krankenhaus der Barmherzigen Bruder, Trier
- Israel (2):
  - Rambam - Health Care Campus, Haifa
  - Sheba Medical Center Hospital, Ramat Gan
- United Kingdom (5):
  - Papworth Hospital, Papworth Everard, Cambridge
  - Blackpool Victoria Hospital, Blackpool
  - University Hospitals Bristol, Bristol
  - The John Radcliffe Hospital, Oxford
  - University Hospital Southampton, Southampton

REFERENCES:
- [Derived] Amin S, Werner RS, Madsen PL, Krasopoulos G, Taggart DP. Influence of external stenting on venous graft flow parameters in coronary artery bypass grafting: a randomized study. Interact Cardiovasc Thorac Surg. 2018 Jun 1;26(6):926-931. doi: 10.1093/icvts/ivy007. PMID 29373645